CLINICAL TRIAL: NCT00578136
Title: A Randomized-Double Blinded Trial Comparing the Analgesic Efficacy and Side Effects of Rectus Sheath Block vs. Infiltration of Surgical Site for Post Operative Pain Control After Umbilical Hernia Repair Surgery
Brief Title: Analgesic Efficacy After Umbilical Hernia Repair in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Children's Anesthesiology Associates, Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 2006-10-4980
Record Dates: First submitted 2007-12-18; First posted 2007-12-20 (Estimated); Results first posted 2014-08-15 (Estimated); Last update posted 2014-08-15 (Estimated); Status verified 2014-07

CONDITIONS: Umbilical Hernia
Keywords: Rectus Sheath; Local infiltration; Pain Control
MeSH Terms: conditions — Hernia, Umbilical; Agnosia | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): 1) One group will receive the rectus sheath block prior to Umbilical hernia repair.
  Interventions: Drug: Bupivacaine
- 2 (Active Comparator): 2) The second group will receive local anesthetic infiltration of the surgical site at the end the umbilical hernia repair.
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Bupivacaine — Bupivacaine, 0.25%, dose amount is weight based, injection is divided per dise with rectus sheath injection or with local infiltration of the operative area.

SUMMARY:
Umbilical hernia repair is a common painful outpatient procedure performed in children. Often analgesia for this procedure is provided by using local infiltration of the surgical site by the surgeons and perioperative opioids and NSAIDS both IV and orally. The use of opioids can cause adverse side effects which include, but are not limited to nausea, vomiting, itching, and respiratory depression, etc. The rectus sheath block can be performed in these patients to decrease their post operative pain.

DETAILED DESCRIPTION:
Umbilical hernia repair, a common Day Surgery procedure in children, is associated with considerable postoperative discomfort. The patient has to meet certain discharge criteria such as tolerating liquids, adequate level of analgesia, etc., prior to being discharged from the day surgery unit.

Currently, both rectus sheath block and local infiltration of the surgical site are used for providing post-operative analgesia for umbilical hernia repair surgery. The local infiltration can only be done at the end of the surgical procedure as it could alter the planes of the surgical field if performed preoperatively. We believe that the analgesia provided prior to the surgical incision will decrease the amount of intraoperative and postoperative opioids used and the subsequent side effects of these medications (5,6). The rectus sheath block, a regional anesthetic technique, offers possible improved pain management following umbilical hernia repair in a recent observational study (1-3,7). We will perform a double-blinded, randomized study to compare the efficacy of rectus sheath block and surgical infiltration in providing postoperative analgesia.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects ages > 5 to < 18 years.
2. American Society of Anesthesiology (ASA)physical status 1 or 2.
3. Patients who undergo an umbilical hernia repair at CHOP.

Exclusion Criteria:

1. Parents/patients refusal to the placement of a rectus sheath nerve block.
2. Subjects with allergy to bupivacaine.
3. Patients who are developmentally delayed which precludes their participation in pain scale reporting.
4. Parents who do not comprehend English sufficiently well to read the consent and ask questions.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2006-11; Primary Completion 2009-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harshad Gurnaney, MBBS, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's hospital of Philadelphia, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 52 patients completed the study, having hernia repair as a day-surgery procedure.
Pre-assignment Details: We screened 120 subjects and excluded 66, 35 patients did not fit the criteria and 31 patients declined to participate. 54 subjects were randomized to receive either a rectus sheath block or local anesthetic infiltration. Two randomized subjects did not get the intervention. 52 subjects did get the intervention - 26 in each arm.
Groups:
- Rectus Sheath Block: 1) One group will receive the rectus sheath block prior to Umbilical hernia repair.
- Local Infiltration: 2) The second group will receive local anesthetic infiltration of the surgical site at the end the umbilical hernia repair.
Period: Overall Study
Arm/Group | Rectus Sheath Block | Local Infiltration
Started | 27 | 27
Completed | 26 | 26
Not Completed | 1 | 1
Not completed — Not given intervention | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rectus Sheath Block | Local Infiltration | Total
Number analyzed (Participants) | 26 | 26 | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 26 | 26 | 52
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.7 (.88) | 7.9 (.88) | 7.8 (.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 24
  Male | 14 | 14 | 28
Region of Enrollment [Number; unit: participants]
  United States | 26 | 26 | 52

OUTCOME MEASURES:

1. Primary Outcome: The Amount of Intravenous and Oral Opioids Used by Patients Who Receive a Rectus Sheath Nerve Block and Those Who Receive Local Infiltration of the Surgical Site for Postoperative Analgesia.
Description: total postoperative opioid and any additional analgesic medications.
Time Frame: immediate to 24 hour post-operatively
Measure: Mean (95% Confidence Interval); unit: mg kg-1
Arm/Group | Rectus Sheath Block | Local Infiltration
Number analyzed (Participants) | 26 | 26
mg kg-1 | 0.07 [0.05 to 0.09] | 0.13 [0.09 to 0.17]
Statistical Analysis 1: Comparison: Rectus Sheath Block vs Local Infiltration; Assuming the opioid requirement in the local infiltration group to be 0.2mg kg-1 and in the rectus sheath block group to be 0.1mg kg-1, a sample size of 44 patients (22 in each group) will have a power of 80% to detect a difference in means of 0.1mg kg-1 with a 0.005 two-sided significance level; Test type: Superiority or Other; p = 0.008, Wilcoxon (Mann-Whitney); The Wilcoxon rank-sum test was used because the study did not have a normal distribution using the Kolmogorov-Smirnov test (p<0.01)

2. Secondary Outcome: The Duration of Analgesia Based on Time to First Rescue Med, the Quality of Analgesia Based on Modified FACES Scale, and the Incidence of Side Effects: Nausea, Vomiting, Pruritus, and Assess Patient Satisfaction With Pain Management.
Description: difference in time to rescue analgesic and the differences in side effects for the two groups.
Time Frame: immediate to 24 hours post-operatively
Population: Time to first rescue dose of opioid medication.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Rectus Sheath Block | Local Infiltration
Number analyzed (Participants) | 26 | 26
minutes | 49.70 (36.94) | 32.35 (29.39)

ADVERSE EVENTS:
Arm/Group | Rectus Sheath Block | Local Infiltration
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/26
Other Adverse Events (participants affected / at risk) | 2/26 | 1/26
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rectus Sheath Block (N=26) | Local Infiltration (N=26)
nausea (Gastrointestinal disorders) | 2 (2) | 1 (1)
vomiting (Gastrointestinal disorders) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes